CLINICAL TRIAL: NCT04297683
Title: HEALEY ALS Platform Trial
Brief Title: HEALEY ALS Platform Trial - Master Protocol
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Master Protocol; Lou Gehrig's Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — zilucoplan; pridopidine

STUDY DESIGN:
Intervention Model Description: As new investigational products become available, additional regimens will be added to the HEALEY ALS Platform Trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research participants, care providers, investigators and site staff (i.e. outcome assessors) will not be blinded to the regimen assignment, but they will be blinded to active product or matching placebo assignment and this blind will be maintained throughout the study. Quadruple masking remains consistent across all regimens which may start at different time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Regimen A - Zilucoplan (Experimental): Participants are randomized to receive either active zilucoplan or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: Zilucoplan
- Regimen B - Verdiperstat (Experimental): Participants are randomized to receive either active verdiperstat or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: Verdiperstat
- Regimen C - CNM-Au8 (Experimental): Participants are randomized to receive either active CNM-Au8 or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: CNM-Au8
- Regimen D - Pridopidine (Experimental): Participants are randomized to receive either active Pridopidine or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: Pridopidine
- Regimen E - SLS-005 Trehalose (Experimental): Participants are randomized to receive either active SLS-005 Trehalose or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: SLS-005 Trehalose
- Regimen F- ABBV-CLS-7262 (Experimental): Participants are randomized to receive either active ABBV-CLS-7262 or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: ABBV-CLS-7262
- Regimen G - DNL343 (Experimental): Participants are randomized to receive either active DNL343 or matching placebo.
  NO LONGER RECRUITING; RESULTS REPORTED.
  Interventions: Drug: DNL343
- Regimen I - NUZ-001 (Experimental): Participants are randomized to receive either active NUZ-001 or matching placebo.
  Interventions: Drug: NUZ-001

INTERVENTIONS:
Drug: Zilucoplan — Drug: Zilucoplan Administration: Subcutaneous injection Dose: Minimum of .0.22 mg/kg daily to a maximum dose of 0.42 mg/kg daily, dependent on weight
  Arms: Regimen A - Zilucoplan
Drug: Verdiperstat — Drug: Verdiperstat Administration: Oral Dose: 600mg twice daily
  Arms: Regimen B - Verdiperstat
Drug: CNM-Au8 — Drug: CNM-Au8 Administration: Oral Dose: 30 mg or 60 mg daily
  Arms: Regimen C - CNM-Au8
Drug: Pridopidine — Drug: Pridopidine Administration: Oral Dose: 45mg twice daily
  Arms: Regimen D - Pridopidine
Drug: SLS-005 Trehalose — Drug: SLS-005 Trehalose Administration: Infusion Dose: 0.75 g/kg weekly
  Arms: Regimen E - SLS-005 Trehalose
Drug: ABBV-CLS-7262 — Drug: ABBV-CLS-7162 Administration: Oral Dose: Dose 1 or Dose 2
  Arms: Regimen F- ABBV-CLS-7262
Drug: DNL343 — Drug: DNL343 Administration: Oral Dose: Once per day
  Arms: Regimen G - DNL343
Drug: NUZ-001 — Drug: NUZ-001. Administration: Oral. Dose: Once per day.
  Arms: Regimen I - NUZ-001

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial.

In this trial, multiple investigational products for ALS will be tested simultaneously or sequentially. Each investigational product will be tested in a regimen. Each regimen consists of a placebo-controlled trial, meaning that the active investigational product and matching placebo will be tested in each regimen.

The additional details that govern the testing of each investigational product will be summarized in separate regimen-specific appendices (RSAs). Each regimen will have a separate ClinicalTrials.gov posting, which will include specific information about the regimen. All regimen-specific outcome measures will be detailed in each regimen posting.

Participants will have an equal chance to be randomized to all regimens that are active at the time of screening. Once randomized to a regimen, participants will be randomized in a 3:1 ratio to either study drug or placebo.

The following regimens are active in the trial:

Regimen I - NUZ-001

New regimens will be continuously added as new investigational products become available. The HEALEY ALS Platform Trial will enroll additional participants as each new regimen is available.

ELIGIBILITY:
Inclusion Criteria:

1. Sporadic or familial ALS diagnosed as clinically possible, probable, lab-supported probable, or definite ALS defined by revised El Escorial criteria.
2. Age 18 years or older.
3. Capable of providing informed consent and complying with study procedures, in the SI's opinion.
4. Time since onset of weakness due to ALS ≤ 24 months at the time of the Master Protocol Screening Visit.
5. Vital Capacity ≥ 50% of predicted capacity at the time of the Master Protocol Screening Visit measured by Slow Vital Capacity (SVC), or, if required due to pandemic-related restrictions, Forced Vital Capacity (FVC) measured in person.
6. Participants must either not take riluzole or be on a stable dose of riluzole for ≥ 30 days prior to the Master Protocol Screening Visit.
7. Participants must either not take edaravone or have completed at least one cycle (typically 14 days) of edaravone prior to the Master Protocol Screening Visit.
8. Participants must have the ability to swallow pills and liquids at the time of the Master Protocol Screening Visit and, in the SI's opinion, have the ability to swallow for the duration of the study.
9. Geographically accessible to the site.

Exclusion Criteria:

1. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant, according to SI's judgment (e.g., cardiovascular instability, systemic infection), or clinically significant laboratory abnormality or EKG changes. Clinically significant abnormal liver or kidney function is exclusionary. The following values [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN) or estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73m2] are exclusionary regardless of clinical symptoms.
2. Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent, in the SI's opinion.
3. Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
4. Use of investigational treatments for ALS (off-label use or active participation in a clinical trial) within 5 half-lives (if known) or 30 days (whichever is longer) prior to the Master Protocol Screening Visit.
5. Exposure at any time to any gene therapies under investigation for the treatment of ALS (off-label use or investigational).
6. If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or of child-bearing potential and unwilling to use effective contraception, for the duration of the trial and for 3 months, or as specified in each RSA, after discontinuing study treatment.
7. If male of reproductive capacity, unwilling to use effective contraception for the duration of the trial and for 3 months, or as specified in each RSA, after discontinuing study treatment.
8. Anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study, in the SI's opinion.
9. If a participant is being re-screened, the disqualifying condition has not been resolved, or the mandatory wash-out duration has not occurred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | 36 Weeks
  Change in disease severity as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) total score and survival.

SECONDARY OUTCOMES:
Respiratory Function | 36 Weeks
  Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Survival | 36 Weeks
  Comparison of rate of occurrence between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (74):
- United States (74):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Health, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Forbes Norris MDA/ALS Research Center, California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Nova Southeastern University, Davie, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, North Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health/Corewell Health, Grand Rapids, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, P.C./Somnos Clinical Research, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Columbia University, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest Health Science, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Providence Brain and Spine Institute ALS Center, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Penn State Hershey, Hershey, Pennsylvania
  - Jefferson Weinberg ALS Center, Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Penn, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - UTHSCSA, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Henrico, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Berry JD, Maragakis NJ, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Stommel EW, Chase M, Pothier L, Harkey BA, Yu H, Sherman A, Shefner J, Hall M, Kittle G, Babu S, Andrews J, D'Agostino D, Tustison E, Scirocco E, Giacomelli E, Alameda G, Locatelli E, Ho D, Quick A, Ajroud-Driss S, Katz J, Heitzman D, Appel SH, Shroff S, Felice KJ, Simmons Z, Miller T, Olney N, Weiss MD, Goutman SA, Fernandes JA Jr, Jawdat O, Owegi MA, Foster L, Vu T, Ilieva H, Newman DS, Arcila-Londono X, Jackson C, Ladha S, Heiman-Patterson T, Caress J, Swenson A, Peltier A, Lewis R, Fee D, Elliott M, Bedlack R, Kasarskis EJ, Elman L, Rosenfeld J, Walk D, McIlduff CE, Twydell P, Young E, Johnson K, Rezania K, Goyal NA, Cohen JA, Benatar M, Jones V, Glass J, Shah J, Beydoun SR, Wymer JP, Zilliox L, Nayar S, Pattee GL, Martinez-Thompson J, Rynders A, Evan J, Evan J, Hartford A, Sepassi M, Ho KS, Glanzman R, Greenberg B, Hotchkin MT, Paganoni S, Cudkowicz ME; HEALEY ALS Platform Trial Study Group. CNM-Au8 in Amyotrophic Lateral Sclerosis: The HEALEY ALS Platform Trial. JAMA. 2025 Feb 17;333(13):1138-49. doi: 10.1001/jama.2024.27643. Online ahead of print. PMID 40067821
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Shefner JM, Oskarsson B, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Heiman-Patterson T, Chase M, Pothier L, Harkey BA, Yu H, Sherman AV, Hall M, Kittle G, Berry JD, Babu S, Andrews J, D'Agostino D, Tustison E, Scirocco E, Giacomelli E, Alameda G, Locatelli E, Ho D, Quick A, Ajroud-Driss S, Katz J, Heitzman D, Appel SH, Shroff S, Felice K, Maragakis NJ, Simmons Z, Miller TM, Olney N, Weiss MD, Goutman SA, Fernandes JA, Jawdat O, Owegi MA, Foster LA, Vu T, Ilieva H, Newman DS, Arcila-Londono X, Jackson CE, Ladha S, Caress JB, Swenson A, Peltier A, Lewis RA, Fee D, Elliott M, Bedlack R, Kasarskis EJ, Elman L, Rosenfeld J, Walk D, McIlduff C, Twydell P, Young E, Johnson K, Rezania K, Goyal NA, Cohen JA, Benatar M, Jones V, Shah J, Beydoun SR, Wymer JP, Zilliox L, Nayar S, Pattee GL, Martinez-Thompson J, Leitner ML, Chen K, Goldberg YP, Cohen Y, Geva M, Hayden MR, Paganoni S, Cudkowicz ME; HEALEY ALS Platform Trial Study Group. Pridopidine in Amyotrophic Lateral Sclerosis: The HEALEY ALS Platform Trial. JAMA. 2025 Feb 17;333(13):1128-37. doi: 10.1001/jama.2024.26429. Online ahead of print. PMID 40067755
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Andrews J, Paganoni S, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Young E, Chase M, Pothier L, Harkey B, Yu H, Sherman A, Shefner J, Hall M, Kittle G, Connolly MR, Berry JD, D'Agostino D, Tustison E, Giacomelli E, Scirocco E, Alameda G, Locatelli E, Ho D, Quick A, Heitzman D, Ajroud-Driss S, Appel SH, Shroff S, Katz J, Felice K, Maragakis NJ, Simmons Z, Goutman SA, Olney N, Miller T, Fernandes JA, Ilieva H, Jawdat O, Weiss MD, Foster L, Vu T, Ladha S, Owegi MA, Newman DS, Arcila-Londono X, Jackson CE, Swenson A, Heiman-Patterson T, Caress J, Fee D, Peltier A, Lewis R, Rosenfeld J, Walk D, Johnson K, Elliott M, Kasarskis EJ, Rutkove S, McIlduff CE, Bedlack R, Elman L, Goyal NA, Rezania K, Twydell P, Benatar M, Glass J, Cohen JA, Jones V, Zilliox L, Wymer JP, Beydoun SR, Shah J, Pattee GL, Martinez-Thompson J, Nayar S, Granit V, Donohue M, Grossman K, Campbell DJ, Qureshi IA, Cudkowicz ME, Babu S. Verdiperstat in Amyotrophic Lateral Sclerosis: Results From the Randomized HEALEY ALS Platform Trial. JAMA Neurol. 2025 Apr;82(4):333-343. doi: 10.1001/jamaneurol.2024.5249. Epub 2025 Feb 17. PMID 40067754
- [Derived] Paganoni S, Fournier CN, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Ajroud-Driss S, Chase M, Pothier L, Harkey BA, Yu H, Sherman AV, Shefner JM, Hall M, Kittle G, Berry JD, Babu S, Andrews J, Dagostino D, Tustison E, Giacomelli E, Scirocco E, Alameda G, Locatelli E, Ho D, Quick A, Katz J, Heitzman D, Appel SH, Shroff S, Felice K, Maragakis NJ, Simmons Z, Miller TM, Olney N, Weiss MD, Goutman SA, Fernandes JA, Jawdat O, Owegi MA, Foster LA, Vu T, Ilieva H, Newman DS, Arcila-Londono X, Jackson CE, Ladha S, Heiman-Patterson T, Caress JB, Swenson A, Peltier A, Lewis R, Fee D, Elliott M, Bedlack R, Kasarskis EJ, Elman L, Rosenfeld J, Walk D, McIlduff C, Twydell P, Young E, Johnson K, Rezania K, Goyal NA, Cohen JA, Benatar M, Jones V, Glass J, Shah J, Beydoun SR, Wymer JP, Zilliox L, Nayar S, Pattee GL, Martinez-Thompson J, Harvey B, Patel S, Mahoney P, Duda PW, Cudkowicz ME; HEALEY ALS Platform Trial Study Group. Efficacy and Safety of Zilucoplan in Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459058. doi: 10.1001/jamanetworkopen.2024.59058. PMID 39960672

DOCUMENTS (1):
  • Study Protocol (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT04297683/Prot_000.pdf